CLINICAL TRIAL: NCT00756301
Title: Cutaneous Administration of Local Anesthetic for Spine Injection Procedures: A Prospective Randomized Controlled Trial of Patient Preferred Method
Brief Title: Cutaneous Administration of Local Anesthetic for Spine Injection Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HUM00002610; 16893
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Spinal Diseases
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Traditional Technique (Active Comparator): Local anesthetic (Lidocaine) injected using traditional technique (involves injecting Lidocaine into the skin first, then into the deeper tissues).
  Interventions: Other: Lidocaine local anesthesia- Alternative
- Alternative Technique (Experimental): Local anesthetic (Lidocaine) injected using an alternative technique (inserting the numbing needle into the deeper tissues first and injecting numbing medication from there up to the skin).
  Interventions: Other: Lidocaine local anesthesia- Alternative
- No Anesthetic (No Intervention): No local anesthetic is used.

INTERVENTIONS:
Other: Lidocaine local anesthesia- Alternative — Local anesthetic (Lidocaine) injected using traditional technique (involves injecting Lidocaine into the skin first, then into the deeper tissues).
  Arms: Alternative Technique; Traditional Technique

SUMMARY:
Interventional spine procedures are an increasingly popular means of diagnosis and treatment of spine disease. By convention, local anesthetics are used at the beginning of these procedures with the goal of minimizing pain. However, the infiltration of the local anesthetic is painful. This initial painful stimulus can heighten pain awareness and cause anxiety or excessive movement during the procedure.

The purpose of this study is to determine patient discomfort with administration of cutaneous local anesthetic prior to interventional spine procedures compared to no anesthetic administration for different gauge procedural needles. Another purpose is to determine patient discomfort with administration of local anesthetic by traditional technique compared to an alternative technique and to develop a standardized technique and criteria for local anesthetic administration during spine injection procedures that minimizes patient pain, and may help reduce the overall risk of these procedures.

We plan to enroll a total of 200-300 subjects coming to Stanford for symmetric bilateral single injections.

DETAILED DESCRIPTION:
Any patient referred by their treating physician for symmetric bilateral single injections (for example, bilateral transforaminal epidural injections, bilateral facet injections, or bilateral SI joint injections, etc.) will provide written informed consent before the procedure is conducted.

The contents of the consent forms will be used to explain the study to patients. Patients with pregnancy, coagulopathy, systemic infection, allergy to contrast dye, mentally disabled or those whom are unable to give informed consent will be excluded from the study.

Three different cutaneous local anesthetic techniques will be investigated, hereafter referred to as (a), (b), and (c), and described in detail here:

1. Local anesthetic injected with a 27-gauge 1.25" needle using traditional technique- formation of a subcutaneous wheal with 0.25cc 1% Lidocaine, then 0.75cc 1% Lidocaine injected along the planned needle trajectory to the hub depth of the 27-gauge needle.
2. Local anesthetic injected with a 27-gauge 1.25" needle using an alternative technique- needle is immediately inserted in the planned needle trajectory to the hub depth. Then 1cc 1% Lidocaine is injected slowly as the needle is withdrawn to the skin creating a small point wheal at the skin prior to removal of the needle.
3. No local anesthetic is used.

   1. Patients are randomly assigned to receive one of three possible combinations of anesthetic techniques (one on each side i.e. (a) & (b), (a) &(c), (b)&(c). Randomized assignment will occur on a rotating basis, i.e.; patient #1 will receive (a)&(b), patient #2 will receive (a)&(c), patient #3 will receive (b)&(c), and so on. Regardless of technique (a), (b), or (c), the following four steps are followed.
   2. After the starting point of the procedure is identified, before placement of any needles, we ask the patient to take note of any subsequent discomfort or pain.
   3. Complete the designated anesthesia technique.
   4. Next, place the treatment needle to a depth of 1 inch. Needle size is determined by the injectionist at the time of the procedure, based on what is determined to be best suited for the patient and the procedure from the following quinke point needles: 26-gauge 3.5", 25-gauge 3.5", or 22-gauge 3.5" needle. The same size needle will be used on each side.
   5. Finally, we ask the patient to rate on a 10 point verbal analog scale the amount of pain they experienced during this time.
   6. Repeat steps 2 thru 5 for the second side of the procedure.

All data is collected during the procedure. There will be no follow-up visits after the procedure.

ELIGIBILITY:
Inclusion Criteria:1. Any patients referred by their treating physician for symmetric bilateral single injections (for example, bilateral transforaminal epidural injections, bilateral facet injections, or bilateral SI joint injections, etc.).

2.Ability to give informed consent. Exclusion Criteria:1.Pregnancy 2.Coagulopathy 3.Systemic infection 4.Allergy to contrast dye 5.Mentally disabled or those whom are unable to give informed consent 6.Those whom are unable to give informed consent in English 7.Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-06; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Pain related to cutaneous anesthesia method | At the time of the injection

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Smuck, Principal Investigator — Stanford University
Locations (1):
- Stanford Univiersity, Redwood City, California, United States